CLINICAL TRIAL: NCT00318981
Title: Efficacy of Concerta in Treating ADHD in Mothers of Children With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry); Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IIS-2003-023
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Adult ADHD
Keywords: Medication trial; ADHD; Concerta; Efficacy trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

INTERVENTIONS:
Drug: Concerta

SUMMARY:
This study involves a 7 week dose-response trial of Concerta™ methylphenidate for mothers of children with ADHD who have ADHD themselves. The aim of this study is to assess the efficacy of Concerta™ in improving adult ADHD symptoms and impairments (primary outcome), as well as observed and reported parenting (secondary outcome). The researchers hypothesize that Concerta™ will significantly decrease mothers ADHD symptoms and impairment, as well as improve observed and reported parenting

DETAILED DESCRIPTION:
There is evidence to suggest that ADHD persists in approximately 50-65% of individuals diagnosed with the disorder during childhood. Due to the familial nature and presumed genetic etiology of this disorder, parents with ADHD are more likely to have children also diagnosed with ADHD. Accordingly, higher rates of adult ADHD have been found in parents of children with ADHD. Recent research has determined that among children with ADHD, there is a 23 times greater rate of ADHD in mothers and a 4 times greater rate of ADHD in fathers relative to parents of children without the disorder.

Research has also suggested that ADHD symptoms that persist into adulthood are impairing in many areas of an individual's life, including their family functioning and work functioning. Spouses of ADHD adults report that their partners' difficulties with communication, task completion, and time management negatively impact their marriages. Similarly, adult ADHD may interfere with parenting in that parents with ADHD may have trouble maintaining their attention during interactions with their children or may overreact to their children's tantrums. However, the role of parents for children with ADHD is critical. Parents of children with ADHD both assist in the delivery of pharmacological and behavioral treatments their children. Therefore, a parent's own ADHD symptoms may interfere with their ability to deliver these vital resources to their child.

Despite this research, little research has been conducted looking at effects of using stimulant medication to treat parents with ADHD who have children with ADHD. In fact, only one case study has examined the effects of treatment for parental ADHD on child treatment response.

The current study seeks to examine the effect of a long-acting stimulant medication (Concerta) on mothers with ADHD who have children with ADHD. Mothers and children receive a free comprehensive ADHD assessment and mothers receive a free 7 week treatment of Concerta under the supervision of a physician.

ELIGIBILITY:
Inclusion Criteria:

Mother:

* Have ADHD or problems paying attention and concentration themselves
* Have a child 6-12 years old with ADHD or possible ADHD
* Be the child's biological mother

Exclusion Criteria:

* Any CURRENT Axis I disorder (including major depression, psychosis, and substance use disorders) but with the exception of minor depressive or anxiety disorders
* Use of Anti-depressant medication
* Mothers with severe tics or Tourette's syndrome, a history of seizures or abnormal EEGs, high blood pressure, or narrowing or blockage of the GI tract
* Any women pregnant or brest-feeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2004-12; Study Completion 2006-12

PRIMARY OUTCOMES:
Adult ADHD symptoms (Conners Adult ADHD Rating Scale)
Impairment ratings (CGI)
Side Effects (Pittsburgh Side Effect Scale)

SECONDARY OUTCOMES:
Parenting measures (Parenting Stress Index, Alabama Parenting Questionnaire, O'Leary Parenting Scale, Observed Parent Child Interaction)

CONTACTS AND LOCATIONS:
Overall Officials: Andre M Chronis, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Children's National Medical Center Regional Outpatient Center, Fairfax, Virginia, United States

REFERENCES:
- [Derived] Chronis-Tuscano A, Seymour KE, Stein MA, Jones HA, Jiles CD, Rooney ME, Conlon CJ, Efron LA, Wagner SA, Pian J, Robb AS. Efficacy of osmotic-release oral system (OROS) methylphenidate for mothers with attention-deficit/hyperactivity disorder (ADHD): preliminary report of effects on ADHD symptoms and parenting. J Clin Psychiatry. 2008 Dec;69(12):1938-47. doi: 10.4088/jcp.v69n1213. Epub 2008 Dec 2. PMID 19192455